CLINICAL TRIAL: NCT06678191
Title: Effectiveness of BDP/FF/G 172/5/9 Fixed Triple Combination on Symptom Scores in Asthma Patients After 6 Months Treatment
Brief Title: Investigation of Fixed Triple Inhaled Combination in Asthmatic Patients, in a Real-life Setting
Acronym: STRENGTH
Status: Recruiting | Type: Observational
Sponsor: Chiesi Hungary Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CHMED_2024/01
Record Dates: First submitted 2024-10-09; First posted 2024-11-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Asthma, Chronic Obstructive Pulmonary Disease (COPD); Asthma Bronchiale
Keywords: Asthma therapy; Fixed triple inhalation treatment; Trimbow
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Glycopyrrolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthmatic patients switched to Trimbow (BDP/FF/G 172/5/9 μg): Asthmatic patients who had been switched to BDP/FF/G 172/5/9 μg before study enrollment, due to uncontrolled asthma.
  Interventions: Drug: BDP/FF/G (Beclomethasone diprprionate, formoterol fumarate, glycopyrronium bromide) 172/5/9 μg

INTERVENTIONS:
Drug: BDP/FF/G (Beclomethasone diprprionate, formoterol fumarate, glycopyrronium bromide) 172/5/9 μg — In accordance with the requirements of non-interventional studies, the assignment of patients to Trimbow 172/5/9 μg pMDI therapy should be made independently of the study, and patients should only be considered for inclusion in the study after a prior therapeutic decision has been made by a pulmonologist.

SUMMARY:
The mainstay of asthma treatment are ICSs, mostly combined with LABA. In the past decade LAMA had been accepted as an add-on treatment for patients on GINA treatment Steps 4 and 5. Recently, RCTs proved the efficacy and safety of fixed triple combinations of moderate and high dose of ICS and LABA, LAMA in a very selected asthmatic population, resulting in the market authorisation of these products. However, there is a lack of evidence on the real-world effectiveness of these therapies, especially with regards to improvement in symptom scores and quality of life. Also, there is scarcity of data regarding the phenotypes of asthmatics who benefit the most from the use of fixed triple combinations.

DETAILED DESCRIPTION:
Study design Multicentre, national, non-interventional, prospective study evaluating the effectiveness of Trimbow 172/5/9 μg pMDI on symptom scores in 6 months after switch from previous LABA-high dose ICS containing treatment in asthmatics.

Dosage regimen and administration Name of the product: Trimbow 172 micrograms/5 micrograms/9 micrograms pressurised inhalation, solution (henceforth abbreviated as Trimbow 172/5/9 μg pMDI). Each delivered dose (the dose leaving the mouthpiece) contains 172 μg of beclometasone dipropionate, 5 μg of formoterol fumarate dihydrate and 9 μg of glycopyrronium (as 11 μg glycopyrronium bromide). Each metered dose (the dose leaving the valve) contains 200 μg of beclometasone dipropionate, 6 μg of formoterol fumarate dihydrate and 10 μg of glycopyrronium (as 12.5 μg glycopyrronium bromide). The recommended dose is two inhalations twice daily. The maximum dose is two inhalations twice daily.

1. Aim of the study (research objective)

   Primary objective:

   The main objective is to assess the effectiveness of BDP/FF/G 172/5/9 μg fixed triple combination in a real-world setting, with regards to improvements in symptom scores (ACT).
2. Test sample and method, recruitment principle No patient recruitment will be performed. Eligible patients will be enrolled during the participating physicians' regular asthma patient management and patients' written informed consent. Patient inclusion will take place among patients having severe asthma and attending pulmonology outpatient clinics (the chosen study sites are attached as annexes to the study protocol), strictly at the time of the patients' visit. The planned number of patients is 800.
3. Structure of the study In accordance with the requirements of non-interventional studies, the assignment of patients to Trimbow 172/5/9 μg pMDI therapy should be made independently of the study, and patients should only be considered for inclusion in the study after a prior therapeutic decision has been made by a pulmonologist. Patient enrolment can take place after the patient has been fully informed about the purpose of the study and all of its details, and the patient has read and signed the patient information leaflet and patient consent form, including any questions they may have. Once this has taken place, the data that would have been generated anyway during the outpatient examination of the patient in accordance with daily practice can be recorded. This is considered the first visit of the study (Visit 1). During this visit, the patient's main demographic data, information on comorbidities and concomitant medications, previous and current asthma therapies, asthma specific assessment (including ACT), exacerbation history, post-dose lung function values (if spirometry data is available), laboratory results (if a laboratory test is performed during the visit or was performed recently), results of other medical examinations (e.g., chest X-ray) if performed regardless of the study, maintenance and reliever inhaled & non-inhaled therapies (former and new) baseline quality of life based on the asthma quality of life (EQ-5D-5L) questionnaire, and adherence to therapy based on Test of Adherence to Inhalers® (TAI-12) questionnaire are recorded. Patients will then attend two additional visits 30 days and 6 months after enrolment as per routine clinical practice (Visits 2 and 3). During these visits, data will also be recorded, once again, according to routine clinical practice. Assessing the usage of rescue medications and patient adherence are also planned with the use of electronic health record system (EESZT)-verified prescription dispensations (optional for investigators). Visit 4 will be a long-term follow-up to assess the exploratory endpoint of exacerbations rates.

   If the patient's maintenance therapy changes during the study as decided by the treating pulmonologist, and the patient is no longer receiving Trimbow 172/5/9 μg pMDI, the patient will be automatically excluded from this NIS. The fact of the therapy modification and its exact date must be recorded on the "current medication" form in the eCRF (electronic Case Report Form) of the next visit. If the change in therapy is related to a suspected adverse reaction, it should be reported separately on the eCRF platform in accordance with section 9 of this protocol ('Collection, recording and reporting of medication safety data').

   This NIS is open to all eligible patients according to the inclusion and exclusion criteria. Permitted concomitant treatments: allowed all medications according to local clinical practice (any non-inhalation therapy for asthma or other diseases) and reliever (short-acting bronchodilators) inhaled therapies for asthma. The data to be recorded will be detailed in the study data sheet that forms part of the protocol. The data is recorded in the eCRF (MrAgent - Medisol Development Ltd., see also at 10.1.) system, with consideration to the current professional and legal regulations.
4. Start and duration of the study The first patient enrolment will take place after receiving approval from the National Public Health Center (NPHC), based on a beneficial assessment of the Medical Research Council of Hungary. The study is planned to start on September 16, 2024. Accordingly, first patient first visit (FPFV) is also planned to take place in September, 2024. The launch of the participating centres is planned in two waves, in the autumn of 2024 and in the spring of 2025. Each centre will have 12 months to enrol patients. After the last visit of the last patient (LPLV), centres will have one month to collect all missing data / correct any data flagged as queries during monitoring. Thus, the LPLV will take place on Oct 31, 2026 (primary endpoint) and 30 April, 2027 (exploratory endpoint), respectively. The study is planned to be concluded on August 31, 2027.
5. Data to be recorded during the visits A total of 4 visits will be performed for the assessment of the primary and secondary endpoints during the study. The table below summarises the data collection to be carried out during the visits separately. The patient may be enrolled in the study and their data may only be recorded, if these data would also have been recorded in accordance with standard medical practice.

   * Visit 1: Time of enrolment - a normal visit, according to routine clinical practice. Informed consent and baseline patient characteristics will be collected.
   * Visit 2: 1 month after enrolment (± 2-3 workdays)
   * Visit 3: 6 months after enrolment (± 5-7 workdays)
   * Visit 4: 12 months after enrolment (± 10-15 days)

ELIGIBILITY:
INCLUSION CRITERIA:

* Physician-confirmed clinical diagnosis of asthma according to GINA guidelines and treated for at least 3 years before inclusion
* Patients ≥ 18 years of age in ambulatory care
* Uncontrolled asthma according to the physician's clinical assessment despite the use of

  1. LABA - high dose ICS OR
  2. LABA - high-dose ICS + LAMA multi-inhaler triple therapy for a minimum of three months.
* Patients who are eligible for the use of Trimbow 172/5/9 μg pMDI according to the SmPC and the financing protocol for asthma

  1. At least on exacerbation, requiring systemic (oral or intravenous) corticosteroids in the previous 12 months
  2. Uncontrolled asthma (ACT≤15)
  3. FEV1<80% at baseline
* Inhaled asthma therapy was changed to Trimbow 172/5/9 μg pMDI no more than 1 week prior to OR on the day of study inclusion
* Patient provided written, informed consent to study participation

EXCLUSION CRITERIA:

* Participation in any clinical trial within 30 days prior to enrolment
* Patients hospitalized due to an exacerbation of their asthma within the last 4 weeks prior to enrolment
* Another respiratory condition, apart from asthma or COPD, that may interfere with the effectiveness of the treatment studied AND/OR another important clinical situation that may interfere with patient's compliance with the treatment.
* Continuous use of oral (>5 mg prednisolone/day OR >4 mg methylprednisolone/day) OR intravenous corticosteroids CHMED_2024/01 Prof. Dr. Lilla Tamási 8(17)
* Use of continuous oxygen therapy
* Any malignant disease in the last 5 years
* Tuberculosis (active or anamnestic)
* Actual or previous use of biologics for asthma treatment in the past 12 months
* All exclusion criteria listed in Trimbow 172/5/9 μg pMDI SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients treated at GINA step 5, uncontrolled with ICS-LABA, containing high dose ICS.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Asthma control Test | 6 months
  Change (improvement) of asthma control test (ACT) score, during the 6 months of treatment (Visit 3), compared to the score at baseline.
Asthma control Test 2 | 6 months
  • The percentage of patients achieving an improvement in asthma control test (ACT) score of 3 points (MCID, minimum clinically important difference) or more, after the 6 months treatment (Visit 3) compared to baseline.

SECONDARY OUTCOMES:
Asthma control test change | 6 months
  The percentage of patients achieving an improvement according to asthma control levels (uncontrolled= ACT ≤15; partially controlled= 15<ACT<20; controlled 20≤ACT)
HRQoL | 6 months
  Change in Health-related QoL was assessed by measuring the 5-level EuroQoL 5-dimension component (EQ-5D-5L) index score at Visit 3 (6 months), compared to the baseline visit 1 (Week 0), regarding the assessment of the impact of Asthma on the patient's quality of life.
Adherence | 6 months
  Change in Test of Adherence to Inhalers® (TAI-12) score at Visit 3 (6 months) compared to baseline visit (Visit 1, week 0) regarding adherence to treatment with use of the Trimbow 172/5/9 μg pMDI.
Lung function | 6 months
  Change in spirometric parameters: FEV1, FVC, FEV1/FVC, at Visit 3 (6 months), compared to the baseline Visit 1 (Week 0), with use of the Trimbow 172/5/9 μg pMDI.

OTHER OUTCOMES:
Exacerbations | 12 months
  Changes in moderate and severe exacerbation rates at Visit 4 (12 months), compared to the baseline Visit 1 (Week 0), with use of the Trimbow 172/5/9 μg pMDI

CONTACTS AND LOCATIONS:
Locations (45):
- Hungary (45):
  - Békés Megyei Központi Kórház, 2. Tüdőgyógyászat szakrendelés - 1. rendelés, Békéscsaba
  - Kispesti Egészségügyi Intézet Tüdőgondozó, Ernyőképszűrő állomás, Budapest
  - Országos Korányi Pulmonológiai Intézet (OKPI), Budapest
  - Semmelweis Egyetem, Általános Orvostudományi Kar, Pulmonológiai Klinika, Budapest
  - Szent Kristóf Szakrendelő XI. Kerületi Tüdőgondozó, Budapest
  - Szent Kristóf Szakrendelő XXII. Kerületi Tüdőgondozó, Budapest
  - XVI. Kerület Kertvárosi Egészségügyi Szolgálata, Tüdőgyógyászat, Budapest
  - Csornai Margit Kórház Tüdőbeteggondozó Intézet, Csorna
  - DE Klinikai Központ, Tüdőgyógyászati Klinika, Debrecen
  - Debreceni Egyetem Kenézy Gyula Egyetemi Kórház Pulmonológiai Részleg, Debrecen
  - Debreceni Egyetem Klinikai Központ Allergológiai Szakrendelés, Debrecen
  - SZTE SZAKK Deszki Multidiszciplináris Centrum, Deszk
  - Dunakeszi-SZTK Nonprofit Kft. Tüdőgyógyászat, Dunakeszi
  - Vaszary Kolos Kórház Tüdőgondozó Esztergom, Esztergom
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Fehérgyarmat
  - Bugát Pál Kórház Tüdőbeteg Gondozó Intézet, Gyöngyös
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Békés Megyei Központi Kórház 1. Tüdőgyógyászat Szakrendelés, Gyula
  - Hajduböszörmény ESZ-V Nonprofit Kft Tüdőgyógyászat, Hajdúböszörmény
  - Tüdőgondozó / Szent Erzsébet Kórház, Jászberény
  - Szent Kereszt Kórház Kalocsa,Tüdőgyógyászati Szakrendelés, Kalocsa
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Keszthelyi Kórház Tüdőgondozó, Keszthely
  - Kisteleki Egészségügyi Központi Nonprofit Kft., Kistelek
  - Szent Damján Görögkatolikus Kórház Tüdőgyógyászati gondozó 1., Kisvárda
  - Selye János Kórház Tüdőgyógyászati Szakellátás, Komárom
  - Kunszentmárton Városi Egészségügyi Központ Tüdőgyógyászat, Kunszentmárton
  - Szaplonczay Manó Marcali Kórház Tüdőgyógyászati Szakrendelés, Marcali
  - Mátrai Gyógyintézet Légzőszervi szakrendelés, Mátraháza
  - Karolina Kórház-Rendelőintézet Mosonmagyaróvár, Mosonmagyaróvár
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Nyírbátor
  - Szabolcs-Szatmár- Bereg Megyei Kórházak és Egyetemi Oktatókórház Megyei-Városi Tüdőgondozó, Nyíregyháza
  - Orosházi Kórház Tüdőgondozó, Orosháza
  - Margit Kórház Pásztó Tüdőgyógyászati Szakrendelés, Pásztó
  - Egyesített Egészségügyi Intézmények Tüdőgondozó, Pécs
  - Sarkadi Kistérségi Járóbeteg Szakellátó Központ, Sarkad
  - Siófoki Kórház-Rendelőintézet Tüdőgondozó, Siófok
  - Csongrád Megyei Mellkasi Betegségek Szakkórháza, Tüdőgondozó Intézet, Szeged
  - Alba Szűrőközpont, Székesfehérvár
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Tüdőbeteg Gondozó, Városkörnyék I. Szakrendelés Székesfehérvár, Székesfehérvár
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelőintézet Tüdőgyógyászati Szakrendelés, Szolnok
  - Markusovszky Egyetemi Oktatókórház, Szombathely
  - Református Pulmonológiai Centrum, Törökbálint, Törökbálint
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg

IPD SHARING:
Plan to Share IPD: No
IDP is sole property of the sponsor and will only be eligible upon reasonable request.